CLINICAL TRIAL: NCT00636857
Title: Postoperative Hyponatremia - Are There Gender Differences?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Moen, Senior Consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKOISR10003
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Hyponatremia
Keywords: Water-Electrolyte Imbalance
MeSH Terms: conditions — Hyponatremia; Water-Electrolyte Imbalance | interventions — Hypodermoclysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Perioperative fluid management based on body weight
  Interventions: Procedure: Fluid administration
- II (Active Comparator): Perioperative fluid management based on Lean Body Mass (LBM)
  Interventions: Procedure: Perioperative fluid management based on Lean Body Mass

INTERVENTIONS:
Procedure: Fluid administration — Preoperative: bolus of 10 ml/kg body weight. During operation: 5 ml/kg body weight/hr. Postoperative: 3 ml/kg body weight/hr
  Other Names: Fluid administration by body weight
  Arms: I
Procedure: Perioperative fluid management based on Lean Body Mass — Preoperative: bolus of 12 ml/kg LBM. During operation: 6 ml/kg LBM/hr. Postoperative: 3.5 ml/kg LBM/hr
  Other Names: Fluid administration by Lean Body Mass
  Arms: II

SUMMARY:
The proposed study will focus on anesthesia and anesthesia-induced hypotension as a possible cause for postoperative fluid retention and hyponatremia, and investigate gender differences in this response.

DETAILED DESCRIPTION:
30 healthy women and 30 healthy men, who are scheduled for surgery of the middle ear or parotic gland are included in the study. Within each gender group, the subjects are randomized to receive perioperative intravenous fluid regimes either based on body weight or lean body mass (LBM). The surgery lasts for at least 3 hours, the intervention period (fluid administration according to protocol) will last 10-12 hours, the study period will be 20-24 hours. Blood samples for analysis of plasma sodium, potassium, glucose and osmolality are collected preoperatively and the following morning together with analysis of urine produced during the study period.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical status I-II
* Subjects scheduled for otorinolaryngoiatric surgery in general anesthesia of at least 3 hours duration

Exclusion Criteria:

* BMI less than 18
* BMI greater than 33
* Diabetes mellitus requiring medication
* Treatment with diuretics
* ACE-inhibitors
* Angiotensin II antagonists
* Cortisone
* Lithium
* Diseases of the kidney
* Females:

  * Pregnancy
  * Menopause
  * Endocrine dysfunction influencing menstruation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change between preoperative and postoperative plasma sodium concentration | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ullman, MD., PhD., Principal Investigator — Dept of Anesthesia and Intensive Care, Karolinska University Hospital, Stockholm,
Locations (5):
- Sweden (5):
  - Department of Anesthesia and Intensive Care, Karolinska University Hospital Huddinge, Stockholm, Stockholm County
  - Dept of Anaesthesia and Intensive Care, Kalmar County Hospital, Kalmar
  - Department of Anaesthesia and Operation, Linköping
  - Dept. of Anesthesiology and Intensive Care, Karolinska University Hospital, Solna, Stockholm
  - Dept of Anaesthesia and Intensive Care, Uppsala University Hospital, Uppsala